CLINICAL TRIAL: NCT03642132
Title: A RANDOMIZED, OPEN-LABEL, MULTICENTER, PHASE 3 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF AVELUMAB IN COMBINATION WITH CHEMOTHERAPY FOLLOWED BY MAINTENANCE THERAPY OF AVELUMAB IN COMBINATION WITH THE POLY (ADENOSINE DIPHOSPHATE [ADP]-RIBOSE) POLYMERASE (PARP) INHIBITOR TALAZOPARIB IN PATIENTS WITH PREVIOUSLY UNTREATED ADVANCED OVARIAN CANCER (JAVELIN OVARIAN PARP100)
Brief Title: Avelumab and Talazoparib in Untreated Advanced Ovarian Cancer (JAVELIN OVARIAN PARP 100)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Phase 3 B9991010 study was stopped due to futility of efficacy at interim analysis on 21Dec2018, and approvals of PARP inhibitors in front-line maintenance setting, Pfizer decided stopping enrollment in the B9991030 study on 19Mar2019.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991030; 2017-004456-30 (EudraCT Number); B9991030 (Other: Alias Study Number); JAVELIN OVARIAN PARP 100 (Other: Alias Study Number)
Record Dates: First submitted 2018-07-13; First posted 2018-08-22 (Actual); Results first posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: untreated epithelial ovarian cancer; fallopian tube cancer; primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Drug Therapy; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- chemotherapy, avelumab and talazoparib (Experimental): Platinum-based chemotherapy + avelumab followed by avelumab + talazoparib maintenance
  Interventions: Drug: Chemotherapy + avelumab followed by avelumab + talazoparib
- chemotherapy, and talazoparib (Experimental): Platinum-based chemotherapy followed by talazoparib maintenance
  Interventions: Drug: Chemotherapy followed by talazoparib maintenance
- chemotherapy and bevacizumab (Active Comparator): Platinum-based chemotherapy + bevacizumab followed by bevacizumab maintenance
  Interventions: Drug: Chemotherapy + bevacizumab followed by bevacizumab

INTERVENTIONS:
Drug: Chemotherapy + avelumab followed by avelumab + talazoparib — Chemotherapy Period Paclitaxel Carboplatin Avelumab
  Maintenance Period Avelumab Talazoparib
  Arms: chemotherapy, avelumab and talazoparib
Drug: Chemotherapy followed by talazoparib maintenance — Chemotherapy Period Paclitaxel Carboplatin
  Maintenance Period Talazoparib
  Arms: chemotherapy, and talazoparib
Drug: Chemotherapy + bevacizumab followed by bevacizumab — Chemotherapy Period Paclitaxel Carboplatin Bevacizumab
  Maintenance Period Bevacizumab
  Arms: chemotherapy and bevacizumab

SUMMARY:
JAVELIN Ovarian PARP 100 (B9991030) is an open-label, randomized study designed to evaluate the efficacy and safety of avelumab in combination with chemotherapy followed by maintenance therapy of avelumab in combination with talazoparib versus an active comparator in treatment-naïve patients with locally advanced or metastatic ovarian cancer (Stage III or Stage IV). On March 19, 2019, Sponsors alliance announced the discontinuation of the ongoing Phase III study, and the decision was based on several factors, including previous announced interim results from JAVELIN Ovarian 100 study (B9991010). Patients who remain in B9991030 study will continue receiving their randomized treatment assigned and will be monitored for appropriate safety assessments until treatment discontinuation.

DETAILED DESCRIPTION:
JAVELIN Ovarian PARP 100 (B9991030) is an open-label, international, multi-center, randomized study designed to evaluate the efficacy and safety of avelumab in combination with chemotherapy followed by maintenance therapy of avelumab in combination with talazoparib versus an active comparator in treatment-naïve patients with locally advanced or metastatic ovarian cancer (Stage III or Stage IV). The primary endpoint is progression-free survival (PFS) as determined based on blinded independent central review (BICR) assessment per RECIST v1.1.

On March 19, 2019, Sponsors alliance announced the discontinuation of the ongoing Phase III JAVELIN Ovarian PARP 100 study. The alliance has notified health authorities and trial investigators of the decision to discontinue the trial. The decision was based on several emerging factors since the trial's initiation, including the previously announced interim results from JAVELIN Ovarian 100 study (B9991010), which was stopped due to futility of efficacy at a planned interim analysis on 21 December 2018. The alliance determined that the degree of benefit observed with avelumab in frontline ovarian cancer in that study does not support continuation of the JAVELIN Ovarian PARP 100 trial in an unselected patient population and emphasizes the need to better understand the role of immunotherapy in ovarian cancer. Additional factors include the rapidly changing treatment landscape and the approval of a PARP inhibitor in the frontline maintenance setting. The decision to discontinue the JAVELIN Ovarian PARP 100 trial was not made for safety reasons.

Patients who remain in the study will continue receiving investigational products according to their randomized treatment assignment and will be monitored for appropriate safety assessments until treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage III IV epithelial ovarian, fallopian tube, or primary peritoneal cancer including carcinosarcoma with high-grade serous component.
* Patients must be candidates for bevacizumab in combination with platinum based chemotherapy and previously untreated.
* Must have completed a primary surgical debulking procedure, or be candidates for neoadjuvant chemotherapy with planned interval debulking surgery.

  1. Patients who completed primary debulking must have had incompletely resected disease that is macroscopically/grossly visible and at least with lesions >1 mm and be randomized at a maximum of 8 weeks after surgery.
  2. For patients who are candidates for neoadjuvant chemotherapy, the diagnoses must have been confirmed by:

     * Core tissue (not fine-needle aspiration) biopsy is required for diagnosis.
     * Stage IIIC-IV documented via imaging or surgery (without attempt at cytoreduction).
     * Serum CA-125/CEA ratio >25. If the serum CA-125/CEA ratio is <25, then workup should be negative for the presence of a primary gastrointestinal or breast malignancy (<6 weeks before start of neoadjuvant treatment).
     * Randomization must occur within 8 weeks after diagnosis.
* Availability of an archival FFPE tumor tissue block or a minimum of 25 slides, together with an accompanying original H&E slide. If archived FFPE tissue is not available, a de novo (ie, fresh) tumor sample must be obtained in accordance with local institutional practice for tumor biopsies. Tumor tissue must contain 40% or greater tumor nuclei per central laboratory assessment.
* ECOG performance status 0-1
* Age >=18 years (or >=20 years in Japan).
* Adequate bone marrow, hepatic, and renal function and blood coagulation

Exclusion Criteria:

* Non-epithelial tumors or ovarian tumors with low malignant potential (ie, borderline tumors) or mucinous tumors.
* Patients for whom intraperitoneal cytotoxic chemotherapy is planned.
* Prior exposure to immunotherapy with interleukin (IL)-2, interferon alpha (IFN-α), or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte associated antigen 4 (anti-CTLA4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, excluding therapeutic anticancer vaccines.
* Prior treatment with a PARP inhibitor.
* Prior treatment with any anti-vascular endothelial growth factor (VEGF) drug, including bevacizumab.
* Major surgery (other than debulking or exploratory surgery for ovarian cancer) for any reason within 4 weeks prior to randomization and/or incomplete recovery from surgery.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Prior targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their ovarian, peritoneal primary or fallopian tube carcinoma.
* Prior organ transplantation including allogenic stem cell transplantation.
* Diagnosis of Myelodysplastic Syndrome (MDS).
* Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (37):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Sansum Clinic, Santa Barbara, California
  - Sansum Clinic, Solvang, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - NYU Winthrop Hospital, Gynecologic Oncology, Mineola, New York
  - NYU Winthrop Hospital, Infusion Center, Mineola, New York
  - NYU Winthrop Radiology, Mineola, New York
  - Montefiore Medical Center - EPC, The Bronx, New York
  - Montefiore Medical Center, Department of Obstetrics and Gynecology and Women's Health, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center-Centennial Facility, The Bronx, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology, Fort Worth, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - Texas Oncology- San Antonio, San Antonio, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Australia (2):
  - Epworth Foundation trading as Epworth HealthCare, East Melbourne, Victoria
  - Epworth HealthCare, Clinical Trials & Research Centre, Richmond, Victoria
- CHU-UCL Namur/Site Sainte Elisabeth, Namur, Belgium
- Bon Secours Hospital, Cork, Ireland
- Italy (2):
  - Istituto Europeo di Oncologia (IEO), Milan, MI
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM
- Niigata Cancer Center Hospital, Niigata, Japan
- Limited Liability Company "VitaMed" (LLC "VitaMed"), Moscow, Russia
- Singapore (7):
  - Department of Nuclear Medicine and Molecular Imaging, Singapore
  - SingHealth Investigational Medicine Unit, Singapore
  - National Cancer Centre Singapore, Singapore
  - Department of Pathology, Singapore
  - Raffles Hospital, Singapore
  - Raffles Radiology, Singapore
  - Farrer Park Hospital, Singapore
- South Korea (6):
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Clinical Trial Pharmacy, Samsung Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Taipei Veterans General Hospital, Taipei
  - Department of Radiology, Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Division of Pharmacy, Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of 19 March 2019, the sponsor decided to stop enrollment/randomization in the study. A total of 104 participants were screened and 79 participants completed screening and randomized in the study before study discontinuation. As only 11% projected enrollment was met at the time of enrollment stop, the original study endpoints are no longer applicable and/or feasible; only the Safety, PK and Immunogenicity Analysis were done and these data are included in this report.
Groups:
- Chemotherapy +Avelumab -> Avelumab + Talazoparib: In chemotherapy period, participants received paclitaxel 175 mg/m^2 intravenously(IV) over 3 hours followed by carboplatin area under the concentration (AUC) 5 or 6 IV over 15-60 minutes on Days 1 of each 3-week cycle for 6 cycles along with avelumab 800 mg administered IV on Day 1 of each 3-week cycle for 6 cycles.
  In maintenance period, participants received avelumab 800 mg administered IV on Days 1, 15 and 29 of each 6-week cycle in combination with talazoparib 0.75 mg self-administered orally once per day.
  A cycle was defined as 3 weeks (21 days) in the chemotherapy period and 6 weeks (42 days) in the maintenance period, respectively.
- Chemotherapy -> Talazoparib: In chemotherapy period, participants received paclitaxel 175 mg/m^2 IV over 3 hours followed by carboplatin AUC 5 or 6 IV over 15-60 minutes on Days 1 of each 3-week cycle for 6 cycles.
  In maintenance period, participants received talazoparib 0.75 mg self-administered orally once a day, every day of each 6-week cycle.
- Chemotherapy + Bevacizumab -> Bevacizumab: In chemotherapy period, participants received paclitaxel 175 mg/m^2 IV over 3 hours followed by carboplatin AUC 5 or 6 IV over 15-60 minutes on Day 1 of each 3-week cycle for 6 cycles along with bevacizumab 15 mg/kg IV on Day 1 of each 3-week cycle beginning with Cycle 2 for adjuvant participants, and for neoadjuvant participants, bevacizumab was given on Day 1 of each 3-week cycle for Cycles 1, 2, 5, and 6.
  In maintenance period, participants received bevacizumab 15 mg/kg administered IV on Days 1 and 22 of each 6-week cycle.
Period: Chemotherapy Period
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Started | 32 | 13 | 34
Completed | 19 | 8 | 27
Not Completed | 13 | 5 | 7
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Physician's decision | 4 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 3
Not completed — Other | 1 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 3 | 1
Period: Maintenance Period
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Started | 18 | 9 | 23
Completed | 5 | 1 | 9
Not Completed | 13 | 8 | 14
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Physician's decision | 2 | 2 | 2
Not completed — Progressive disease | 9 | 3 | 6
Not completed — Other | 0 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2
Period: Follow-up Period
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Started | 19 | 9 | 28
Completed | 14 | 7 | 24
Not Completed | 5 | 2 | 4
Not completed — Other | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Study terminated by sponsor | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Death | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all randomized participants who received at least 1 dose of study drug (avelumab, talazoparib, bevacizumab, carboplatin, paclitaxel).
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab | Total
Number analyzed (Participants) | 32 | 13 | 34 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.38 (11.32) | 58.46 (12.67) | 63.29 (9.83) | 61.72 (10.93)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 21 | 8 | 20 | 49
  65 =< 75 years | 7 | 4 | 9 | 20
  75 =< 85 years | 4 | 1 | 5 | 10
  >= 85 years | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 13 | 34 | 79
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 5 | 12
  Not Hispanic or Latino | 26 | 11 | 27 | 64
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Blank or African American | 0 | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 3 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 29 | 10 | 24 | 63
  Other | 1 | 0 | 1 | 2
  Unknown | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (On-Treatment Period)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death, was lifethreatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect or considered to be an important medical event. AEs included SAEs and non-serious AEs.
  On-treatment period was defined as the time from the first dose of study treatment through up to 30 days after minimum last dose of study treatment or start day of new anti-cancer drug therapy minus 1 day.
Time Frame: From the first dose of study treatment through up to 30 days after minimum last dose of study treatment or start day of new anti-cancer drug therapy minus 1 day (maximum up to 3.5 years approximately)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug (avelumab, talazoparib, bevacizumab, carboplatin, paclitaxel). Participants was classified according to the study treatment assigned at randomization unless the incorrect treatment(s) was/were received throughout the dosing period in which case participants would be classified according to the first study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 29 | 13 | 34
Participants | 29 | 13 | 34

2. Secondary Outcome: Number of Participants With ADA Against Avelumab by Never and Ever Positive Status
Description: Predose Anti-drug antibodies (ADA) samples were collected within 2 hours prior to avelumab dosing and drawn from the contralateral arm of the avelumab infusion.
Time Frame: Day 1 pre-dose of Cycles 1, 2, 3, and 4 in the chemotherapy period and Days 1 and 29 of Cycle 1 and Day 1 of Cycles 2, 4, 6, and 10 in the maintenance period and at the end of treatment/withdrawal, up to 27 months.
Population: The immunogenicity analysis set was a subset of the safety analysis set and included participants in Arm A (Chemotherapy +Avelumab -> Avelumab + Talazoparib) only, who had at least 1 ADA sample collected. Only avelumab containing arm (Arm A) was included as the analysis was against avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib
Number analyzed (Participants) | 29
Participants
  ADA never-positive | 17
  ADA ever-positive | 12

3. Secondary Outcome: Pre-dose/Trough Concentration (Ctrough) for Avelumab (Chemotherapy Period)
Description: Ctrough was defined as predose concentration during multiple dosing and it was observed directly from data
Time Frame: Day 1 of Cycles 1, 2, 3, and 4 in the chemotherapy period (1 cycle = 3 weeks)
Population: The pharmacokinetic (PK) concentration analysis set was a subset of the safety analysis set and included participants who had at least 1 concentration above the below limit of quantitation (BLQ) of either avelumab or talazoparib. Only avelumab containing arm (Arm A) was applicable as it was an analysis of avelumab concentration. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib
Number analyzed (Participants) | 29
mcg/mL
  Cycle 1 Day 1 0H: number analyzed (Participants) | 28
  Cycle 1 Day 1 0H | 0.000 [0.00 to 5.61]
  Cycle 2 Day 1 0H: number analyzed (Participants) | 23
  Cycle 2 Day 1 0H | 4.370 [0.00 to 10.8]
  Cycle 3 Day 1 0H: number analyzed (Participants) | 19
  Cycle 3 Day 1 0H | 6.100 [0.00 to 20.9]
  Cycle 4 Day 1 0H: number analyzed (Participants) | 9
  Cycle 4 Day 1 0H | 10.00 [0.686 to 16.1]

4. Secondary Outcome: Pre-dose/Trough Concentration (Ctrough) for Avelumab (Maintenance Period)
Description: Ctrough was defined as predose concentration during multiple dosing and it was observed directly from data
Time Frame: Pre-dose on Days 1 and 29 of Cycle 1 and Day 1 of Cycles 2, 4, 6, and 10 in the maintenance period (1 cycle = 6 weeks) and at the end of treatment, up to 27 months.
Population: as for outcome 3
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib
Number analyzed (Participants) | 29
mcg/mL
  Cycle 1 Day 1 0H: number analyzed (Participants) | 16
  Cycle 1 Day 1 0H | 3.470 [0.00 to 25.7]
  Cycle 1 Day 29 0H: number analyzed (Participants) | 15
  Cycle 1 Day 29 0H | 41.60 [19.5 to 78.0]
  Cycle 2 Day 1 0H: number analyzed (Participants) | 8
  Cycle 2 Day 1 0H | 33.90 [25.7 to 63.6]
  Cycle 4 Day 1 0H: number analyzed (Participants) | 3
  Cycle 4 Day 1 0H | 28.60 [23.3 to 41.0]
  Cycle 6 Day 1 0H: number analyzed (Participants) | 1
  Cycle 6 Day 1 0H | 20.6 [20.6 to 20.6]

5. Secondary Outcome: Cmax for Avelumab (Chemotherapy Period)
Description: Cmax was defined as maximum observed plasma concentration and it was observed directly from data
Time Frame: Day 1 of Cycles 1, 2, 3, and 4 in the chemotherapy period (1 cycle = 3 weeks)
Population: as for outcome 3
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib
Number analyzed (Participants) | 29
mcg/mL
  Cycle 1 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 25
  Cycle 1 Day 1 1H/End of infusion(EOI) | 218.0 [132 to 318]
  Cycle 2 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 18
  Cycle 2 Day 1 1H/End of infusion(EOI) | 222.5 [29.8 to 319]
  Cycle 3 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 17
  Cycle 3 Day 1 1H/End of infusion(EOI) | 253.0 [157 to 349]
  Cycle 4 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 19
  Cycle 4 Day 1 1H/End of infusion(EOI) | 243.0 [139 to 343]

6. Secondary Outcome: Cmax for Avelumab (Maintenance Period)
Description: Cmax was defined as maximum observed plasma concentration and it was observed directly from data
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib
Number analyzed (Participants) | 29
mcg/mL
  Cycle 1 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 12
  Cycle 1 Day 1 1H/End of infusion(EOI) | 227.0 [154 to 282]
  Cycle 1 Day 29 1H/End of infusion(EOI): number analyzed (Participants) | 13
  Cycle 1 Day 29 1H/End of infusion(EOI) | 279.0 [190 to 485]
  Cycle 2 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 6
  Cycle 2 Day 1 1H/End of infusion(EOI) | 222.0 [158 to 289]
  Cycle 4 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 2
  Cycle 4 Day 1 1H/End of infusion(EOI) | 225.0 [224 to 226]
  Cycle 6 Day 1 1H/End of infusion(EOI): number analyzed (Participants) | 1
  Cycle 6 Day 1 1H/End of infusion(EOI) | 219.0 [219 to 219]

7. Secondary Outcome: Ctrough for Talazoprib (Maintenance Period)
Description: Ctrough was defined as predose concentration during multiple dosing and it was observed directly from data.
Time Frame: Pre-dose on Days 1, 15 and 29 of Cycle 1
Population: The pharmacokinetic (PK) concentration analysis set was a subset of the safety analysis set and included participants who had at least 1 concentration above the lower limit of quantitation (LLQ) of either avelumab or talazoparib. Only the talazoprib containing arms (Arm A and Arm B) were applicable as it was an analysis of talazoprib concentration. It is anticipated the number of participants for PK concentration analysis set would be different from safety analysis set.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib
Number analyzed (Participants) | 9 | 8
pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 6
  Cycle 1 Day 1 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 | 2425 [1920 to 2930] | 1343 [865 to 1820]
  Cycle 1 Day 29: number analyzed (Participants) | 3 | 3
  Cycle 1 Day 29 | 2500 [2060 to 6470] | 1950 [660 to 3290]

8. Primary Outcome: Progression-free Survival (Participants With Newly Diagnosed Advanced Ovarian Cancer With Defects in DDR+）
Description: Progression-free survival (PFS) was defined as the time from randomization to the date of the first documentation of objective progressive disease (PD) or death due to any cause, whichever occurred first. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm, appearance of one or more new lesions was considered PD.
Time Frame: At screening, 9 and 18 weeks after date of randomization, then every 12 weeks thereafter until PD by Blinded Independent Central Review (BICR) regardless of initiation of new anti-cancer therapy
Population: This OM measure was planned but due to the premature termination of the study and consequent lack of meaningful data, data are not available and no analyses were performed.
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Overall Survival (Participants of Both DDR+ and Unselected DDR Status)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From 9 weeks up to approximately 3.5 years
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Progression-free Survival (Participants of Unselected DDR Status)
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of PD or death due to any cause, whichever occured first.
Time Frame: At screening, 9 and 18 weeks after date of randomization, then every 12 weeks thereafter until PD by BICR regardless of initiation of new anti-cancer therapy, up to approximately 3.5 years.
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Progression-free Survival (Participants of Both DDR+ and Unselected DDR Status)
Description: PFS was defined as the time from randomization to the date of the first documentation of objective progressive disease(PD) or death due to any cause, whichever occured first. Participants was defined as having defective DDR (DDR+) or having intact DDR (DDR ) using a next generation sequencing based assay method.
Time Frame: as for outcome 10
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Progression-free Survival on Next-line Therapy. (Participants of Both DDR+ and Unselected DDR Status)
Description: Progression-free survival on next-line therapy (PFS2) was defined as time from the date of randomization to the start of second subsequent treatment after first documentation of PD, or death from any cause, whichever occured first. Participants was defined as having defective DDR (DDR+) or having intact DDR (DDR ) using a next generation sequencing based assay method
Time Frame: From screening until the participant had objective PD on or prior to start of next-line anti-cancer treatment, and started a second subsequent anti-cancer treatment or the participant died, up to approximately 3.5 years.
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: PFS Per Gynecological Cancer Intergroup Criteria (Participants of Both DDR+ and Unselected DDR Status)
Description: PFS based on investigator assessment per Gynecological Cancer Intergroup criteria (GCIG) would be assessed incorporating both Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and CA 125. Participants was defined as having defective DDR (DDR+) or having intact DDR (DDR ) using a next generation sequencing based assay method.
Time Frame: From screening until death, end of study, or participant withdrawal of consent, whichever occurred first, up to approximately 3.5 years.
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Functional Assessment of Ovarian Symptom Index-18 (FOSI-18) Score
Description: NFOSI-18 was an ovarian cancer-specific symptom index comprised of symptoms rated as highest priority by both oncology clinical experts and women with advanced ovarian cancer. It was specifically designed to be a stand-alone instrument to measure disease-related symptoms, treatment side effects and function/well-being in participants with ovarian cancer.
  The NFOSI-18 has several subscales: disease-related symptoms physical subscale(9 items), disease-related symptoms emotional subscale(1 item), treatment-related side effect subscale (5 items) and functional well-being (3 items). A high score was good. A score of "0" was a severely symptomatic participant and the highest possible score was an asymptomatic participant.
Time Frame: 3 years
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Programmed Death Receptor-1 Ligand-1 (PD-L1) Biomarker Expression in Tumor and Immune Cells as Assessed by Immunohistochemistry (IHC) at Baseline
Description: The number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and inflammatory cells in regions of interest that were defined by tumor cell morphology and the presence or absence of inflammatory cells
Time Frame: Baseline
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Mutations in Key Oncogenes at Baseline
Description: Determination/estimation of the frequency of mutations (total and non-synonymous) present in baseline tumor derived nucleic acid samples and in baseline circulating tumor DNA.
Time Frame: Baseline
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: EuroQol Group 5-Dimension 5-Level (EQ-5D-5L) Score
Description: The EuroQol EQ-5D-5L was a 6 item participant-completed questionnaire designed to assess health status in terms of a single index value or utility score. There are 2 components to the EQ-5D-5L, a Health State Profile which had individuals rate their level of problems (none, slight, moderate, severe, extreme/unable) in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a Visual Analogue Scale (VAS) in which participants rate their overall health status from 0 (worst imaginable) to 100 (best imaginable). Published weights were available that allow for imputation of the index score. Overall index scores ranged from 0 to 1, with low scores representing a higher level of dysfunction.
Time Frame: 3 years
Population: as for outcome 8
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause mortality: collected from the signing of Informed Consent (IC) up to 90 calendar days after the last administration of the investigational product (maximum of approximately 3.5 years). Serious and non-serious adverse events (AEs) were collected from the time of the first dose of study treatment through up to 30 days after last dose of study treatment or the start of new anti-cancer drug therapy minus 1 day (maximum of approximately 3.5 years).
Description: Both non serious AEs and SAEs were recorded on the case report form.
Arm/Group | Chemotherapy +Avelumab -> Avelumab + Talazoparib | Chemotherapy -> Talazoparib | Chemotherapy + Bevacizumab -> Bevacizumab
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/13 | 2/34
Serious Adverse Events (participants affected / at risk) | 9/29 | 4/13 | 15/34
Other Adverse Events (participants affected / at risk) | 29/29 | 13/13 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy +Avelumab -> Avelumab + Talazoparib (N=29) | Chemotherapy -> Talazoparib (N=13) | Chemotherapy + Bevacizumab -> Bevacizumab (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy +Avelumab -> Avelumab + Talazoparib (N=29) | Chemotherapy -> Talazoparib (N=13) | Chemotherapy + Bevacizumab -> Bevacizumab (N=34)
Anaemia (Blood and lymphatic system disorders) | 12 | 3 | 14
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 12 | 5 | 14
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Visual field defect (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 8 | 3 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 1
Constipation (Gastrointestinal disorders) | 9 | 2 | 12
Diarrhoea (Gastrointestinal disorders) | 11 | 3 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 3 | 14
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 4 | 2 | 7
Adverse drug reaction (General disorders) | 0 | 0 | 2
Asthenia (General disorders) | 2 | 3 | 3
Fatigue (General disorders) | 14 | 6 | 9
Gait disturbance (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 4
Pain (General disorders) | 5 | 0 | 2
Peripheral swelling (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 5 | 1 | 4
Temperature intolerance (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 3
Seasonal allergy (Immune system disorders) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 2
Pneumonia (Infections and infestations) | 5 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 1 | 7
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 2 | 2
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3
Amylase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Blood corticotrophin increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 3 | 3
Platelet count decreased (Investigations) | 3 | 0 | 3
Weight increased (Investigations) | 2 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 8 | 4 | 5
Dysgeusia (Nervous system disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 5 | 2 | 10
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 8 | 1 | 12
Paraesthesia (Nervous system disorders) | 1 | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 3
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 2
Taste disorder (Nervous system disorders) | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 3
Depression (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 5 | 2 | 5
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 5 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 11
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 7 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Flushing (Vascular disorders) | 2 | 1 | 3
Hot flush (Vascular disorders) | 3 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 11
Hypotension (Vascular disorders) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
As of 19 March 2019, the sponsor decided to stop enrollment/randomization in the study. A total of 104 participants were screened and 79 participants completed screening and randomized in the study before study discontinuation. As only 11% projected enrollment was met at the time of enrollment stop, the original study endpoints are no longer applicable and/or feasible; only the Safety, PK and Immunogenicity Analysis were done and these data are included in this report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT03642132/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03642132/SAP_001.pdf